CLINICAL TRIAL: NCT03657953
Title: Patient-relevant Outcomes 8 Years After Minimally Invasive Total Hip Replacement - a Randomized Prospective Study
Brief Title: Outcomes 8 Years After Minimal Invasive THA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Stryker Instruments (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THA MIC
Record Dates: First submitted 2018-08-14; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis, Hip
Keywords: Total Hip Arthroplasty; minimally invasive; Patient-relevant outcomes
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: single-center prospective randomized study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- anterior (MI-A) surgical approach (Active Comparator): The minimally invasive anterior surgical approach was carried out using a modified Smith-Petersen access as described by Bender et al. (Bender et al. 2009) with the patient in supine position.
  Interventions: Other: surgical approach
- anterolateral (MI-AL) surgical approach (Active Comparator): For the minimally invasive anterolateral surgical approach, a modified Watson-Jones approach according to Röttinger (Rottinger et al. 2006) was applied with the patient in supine position.
  Interventions: Other: surgical approach
- direct lateral (DLA) surgical approach (Active Comparator): The direct lateral surgical approach was performed according to the technique described by Hardinge et al. (Hardinge et al. 1982) with the patient positioned supine
  Interventions: Other: surgical approach

INTERVENTIONS:
Other: surgical approach

SUMMARY:
There exists only limited scientific evidence concerning medium- to long-term benefits concerning minimally invasive (MI) total hip arthroplasty (THA). The investigators examined in a randomized study design 157 patients 8 years after THA, which were performed via 3 different surgical approaches.

DETAILED DESCRIPTION:
In contrast to reported short-term advantages of minimally invasive (MI) total hip arthroplasty (THA) there exists only limited scientific evidence concerning medium- to long-term benefits.

The investigators therefore sought to answer the following questions: Is the functional medium-term outcome in THA patients with MI-anterior(MI-A) and MI-anterolateral (MI-AL) approach superior to those treated by direct lateral approach (DLA)? Is the level of life quality increased by MI-THA? Is patient satisfaction higher by MI-THA? Is the revision rate reduced by MI-THA?

ELIGIBILITY:
Inclusion Criteria:

* clinical and radiologic signs of advanced hip joint Degeneration
* Patients from age 18 to 75

Exclusion Criteria:

* osteoporosis and
* osteomalacia,
* preceding surgery or radiation therapy in the proximity of the affected hip joint,
* progressive neoplasia,
* preceding or manifest infection of the affected joint and its surrounding soft tissues,
* rheumatoid arthritis,
* hip dysplasia Hartofilakidis type 2 or 3,
* non-compliance,
* chronic neurological or psychiatric diseases,
* ongoing pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Physical function hip - Harris-Hip-Score (HHS) | change from baseline (preoperative) at 8 years after THA
  Harris-Hip-Score (worst=0, best=100)

SECONDARY OUTCOMES:
Physical function hip - WOMAC | change from baseline (preoperative) at 8 years after THA
  WOMAC Total Score (worst=0, best=100)
Satisfaction Level | at 8 years after THA
  Satisfaction scale (worst=0, best=10)
health related Quality of life - Index | change from baseline (preoperative) at 8 years after THA
  EuroQol in 5 dimensions (EQ-5D) Index (worst=0, best=1)
health related Quality of life - VAS | change from baseline (preoperative) at 8 years after THA
  EQ-Visual Analogue Scale (worst=0, best=100)
Physical Activity | change from baseline (preoperative) at 8 years after THA
  University of California, Los Angeles (UCLA) Activity Scale (worst=1, best=10)
Revision rate | at 8 years after THA
  Revision rate using Kaplan-Meier-Survival Analysis
Physical Activity Performance Test: walking | change from baseline (preoperative) at 8 years after THA
  25-meter walking time
Physical Activity Performance Test: stair climbing | change from baseline (preoperative) at 8 years after THA
  5-step walking time

CONTACTS AND LOCATIONS:
Overall Officials: Maik Stiehler, MD, Principal Investigator — University Center for Orthopaedics and Trauma Surgery, University Hospital Carl Gustav
Locations (1):
- University Hospital Dresden, Orthopaedic Department, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No